CLINICAL TRIAL: NCT01875094
Title: Promoting Self-Management in Stroke Survivors Using Health IT
Brief Title: Self-Management in Stroke Survivors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Berman Center for Outcomes and Clinical Research (Other); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1212M25581; R21HS021794 (AHRQ)
Record Dates: First submitted 2013-05-29; First posted 2013-06-11 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-06

CONDITIONS: Stroke; Hypertension
MeSH Terms: conditions — Stroke; Hypertension | interventions — Self-Management

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Self-Management / MTM via Health IT (Experimental): Stroke survivors are trained to measure and enter BP into an online health management tool
  Interventions: Other: Self-Management / MTM using Health IT
- Usual Care (No Intervention)

INTERVENTIONS:
Other: Self-Management / MTM using Health IT
  Arms: Self-Management / MTM via Health IT

SUMMARY:
This is a feasibility study of using health-IT to promote self-management of risk factors in stroke survivors.

ELIGIBILITY:
Inclusion Criteria:

* Acute Stroke Survivors and their caregivers
* English speaking
* History of hypertension

Exclusion Criteria:

-Cannot use the health-IT system

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2012-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Rate of blood pressure control into guideline recommended ranges | 3 months
  The American Heart Association/American Stroke Association (AHA/ASA) have cited the JNC-7 in their guidelines to define normal blood pressure as < 120/80. We will use these guidelines and examine rates (percentage of subjects) of blood pressure control in intervention vs. usual care group.

SECONDARY OUTCOMES:
Medication Compliance | 3 months
  Percent of subjects who have discontinued one or more of the blood pressure medications on their own (i.e. without medical direction) in the intervention vs. usual care group.
Use of online tool | 3 months
  Ease of online health management tool use will be operationalized as the percent of subjects in the intervention group who measure their BP and enter it online at least 75% of the study period, 50% of the study period and those with 25% or less of the study period.

CONTACTS AND LOCATIONS:
Locations (1):
- University_of_Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Lakshminarayan K, Westberg S, Northuis C, Fuller CC, Ikramuddin F, Ezzeddine M, Scherber J, Speedie S. A mHealth-based care model for improving hypertension control in stroke survivors: Pilot RCT. Contemp Clin Trials. 2018 Jul;70:24-34. doi: 10.1016/j.cct.2018.05.005. Epub 2018 May 12. PMID 29763657